CLINICAL TRIAL: NCT07326865
Title: Glucose IV and Its Hepatic Outcomes After a Metabolic Stress Test During Bariatric Surgery in Obese Patients With and Without MASLD
Brief Title: Hepatic Gene Response to Intravenous Glucose in Obese Patients With and Without MASLD Undergoing Bariatric Surgery
Acronym: GHAST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Spaarne Gasthuis (Other)
Responsible Party: Principal Investigator, Max Nieuwdorp, Prof. Dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 2025.0097
Record Dates: First submitted 2025-12-03; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-06

CONDITIONS: MASLD
Keywords: MASLD (Metabolic Associated Steatotic Liver Disease); Obesity; Bariatric surgery; Roux-en-Y gastric bypass (RYGB); [6,6-D2]-labeled glucose; Hepatic gene expression; RNA sequencing; Adipose tissue transcriptomics; Metabolomics; Postprandial metabolism
MeSH Terms: conditions — Obesity | interventions — Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MASLD + Glucose (Experimental): Participants with metabolic associated steatotic liver disease (MASLD) undergoing bariatric surgery receive a 35-gram intravenous bolus of [6,6-D2]-labeled glucose in 150 mL solution.
  Interventions: Other: [6,6-D2]-labeled glucose (intravenous)
- MASLD + Saline (Placebo Comparator): Participants with MASLD undergoing bariatric surgery receive an intravenous infusion of 150 mL saline (0.9% sodium chloride)
  Interventions: Other: Saline (0.9% sodium chloride infusion)
- Non-MASLD + Glucose (Experimental): Participants without MASLD undergoing bariatric surgery receive a 35-gram intravenous bolus of [6,6-D2]-labeled glucose in 150 mL solution.
  Interventions: Other: [6,6-D2]-labeled glucose (intravenous)
- Non-MASLD + Saline (Placebo Comparator): Participants without MASLD undergoing bariatric surgery receive an intravenous infusion of 150 mL saline (0.9% sodium chloride).
  Interventions: Other: Saline (0.9% sodium chloride infusion)

INTERVENTIONS:
Other: [6,6-D2]-labeled glucose (intravenous) — Participants receive a 35-gram intravenous bolus of [6,6-D2]-labeled glucose dissolved in 150 mL solution. The infusion is administered at the start of bariatric surgery over 3-5 minutes via an indwelling catheter. Liver and adipose tissue biopsies are collected before infusion and 45 minutes after infusion to assess transcriptomic changes. Blood samples are taken at multiple timepoints to measure glucose, insulin, and plasma metabolites, metabolites can be traced using the labeled glucose.
  Arms: MASLD + Glucose; Non-MASLD + Glucose
Other: Saline (0.9% sodium chloride infusion) — Participants receive an intravenous infusion of 150 mL saline (0.9% sodium chloride) at the start of bariatric surgery. The infusion is administered over 3-5 minutes via an indwelling catheter. Liver and adipose tissue biopsies are collected before infusion and 45 minutes after infusion to serve as controls for transcriptomic and metabolic changes.
  Other Names: Intravenous saline
  Arms: MASLD + Saline; Non-MASLD + Saline

SUMMARY:
The goal of this clinical trial is to learn how the liver responds to sugar in people with obesity who are having bariatric surgery. Researchers want to understand differences between people with and without metabolic associated steatotic liver disease (MASLD).

The main question is:

Does giving sugar directly into the vein change how liver genes work in people with and without MASLD?

Researchers will compare:

* People with MASLD who receive sugar
* People with MASLD who receive saline (salt water)
* People without MASLD who receive sugar
* People without MASLD who receive saline

During surgery, participants will:

* Receive either a sugar solution (35 grams of glucose in 150 mL fluid) or saline
* Have small samples (biopsies) taken from the liver and fat tissue before and 45 minutes after the infusion
* Provide blood samples to measure sugar, insulin, and other metabolites
* Provide a one-time sample of intestinal tissue that is normally removed during surgery

This study may help explain why MASLD develops and how the liver reacts to sugar. The results could lead to new ways to understand and treat liver disease in people with obesity.

DETAILED DESCRIPTION:
Metabolic Associated Steatotic Liver Disease (MASLD) is the most common chronic liver disease worldwide and a major cause of liver-related illness and death. Current knowledge is largely based on fasting-state liver biopsies, which do not capture the transcriptional changes triggered by nutrient intake. Postprandial dysfunction is a hallmark of MASLD, yet the molecular mechanisms in human liver tissue under metabolic stress remain poorly understood.

This study uses bariatric surgery as a unique opportunity to obtain paired liver and adipose tissue biopsies before and after an intravenous glucose challenge. By administering a 35-gram bolus of [6,6-D2]-labeled glucose during surgery, researchers can mimic the caloric load of a high-sugar meal while controlling for confounding factors such as anesthesia and surgical stress through saline control groups.

The design is a single-center, interventional, 2 × 2 factorial trial with 40 obese participants (20 with MASLD, 20 without MASLD). Participants are randomized to receive either labeled glucose or saline. Biopsies of liver, subcutaneous, omental, and visceral adipose tissue are collected at baseline and 45 minutes after infusion. Jejunal tissue routinely removed during Roux-en-Y gastric bypass is also analyzed for transcriptomic and microbiome profiling.

Primary analyses focus on single-cell RNA sequencing of liver biopsies to identify transcriptional changes induced by glucose infusion and to compare responses between MASLD and non-MASLD participants. Secondary analyses include transcriptomic profiling of adipose depots (subcutaneous, visceral and omental), jejunal tissue, and untargeted metabolomics/proteomics of plasma samples. The use of stable isotope-labeled glucose allows tracing of metabolic pathways, including erythritol synthesis via the pentose phosphate pathway.

This approach builds on prior work done using the BARIA cohort (DOI: 10.1111/joim.13157), which demonstrated that postprandial states reveal clinically relevant differences in metabolic health not apparent in fasting conditions. By integrating tissue transcriptomics, plasma metabolomics, and microbiome data, the GHAST study aims to uncover mechanisms of metabolic dysregulation in MASLD and identify novel therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this study, a subject must meet all of the following criteria:

Adult individuals, age >35 < 65 years old. Stable weight (no more than 3% TWL of initial body weight from screening to surgery) Subjects should be able to give informed consent Subjects agree to have tissue biopsies performed during surgery, that is 2 liver, subcutaneous, visceral and omental biopsies plus a one-time jejunal biopsy.

For obese non-MASLD patients:

* Adult individuals, age >35 < 65 years old.
* BMI ≥ 40 kg/m², or a BMI ≥ 35 kg/m² with an obesity-related comorbidity
* No MASLD based on Fibroscan
* Estimated glomerular filtration rate (eGFR) > 60mL/min/1.73m2

For obese MASLD patients:

* MASLD diagnosis according to Fibroscan
* Compensated liver disease with the following hematologic and biochemical criteria on entry into study:

  * ALAT <10x ULN
  * Hemoglobin > 11g/dL for females and 12 g/dL for males
  * White blood cell (WBC) > 2.5 K/ μL
  * Neutrophil count > 1.5 K μL
  * Platelets > 100 K/μL
  * Total bilirubin <35 μmol/L
  * Albumin >30 g/L
  * TP >80% or INR <1.4
  * Serum creatinine <1.3 mg/dL (men) or <1.1 mg/dL (women) or
* Estimated glomerular filtration rate (eGFR) > 60mL/min/1.73m2

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Use of metformin and SGLT2/ exogenous insulin/GLP-1 RA
* Primary lipid disorder
* Known genetic basis for insulin resistance or glucose intolerance
* All medical and psychiatric conditions except for obesity related diseases.
* Uncontrolled hypertension (RR > 150/95 mmHg)
* Chronic kidney disease (creatinine > 150 umol/L)
* Pregnancy, females who are breastfeeding
* Evidence of another form of liver disease
* History of sustained excess alcohol ingestion: daily consumption >30g/day (3 drinks per day) for males and >20 g/day (2 drinks per day) for females
* Significant systemic or major illnesses other than liver disease, including congestive heart failure (class C and D of the AHA), unstable coronary artery disease, cerebrovascular disease, pulmonary disease, kidney failure, organ transplantation, serious psychiatric disease, active malignancy, compromised immunity
* Body mass index (BMI) >45 kg/m2
* Type 1 or type 2 diabetes
* Hemostasis disorders or current treatment with anticoagulants
* Known heart failure
* Contra-indication for liver biopsy History of/or current cardiac dysrhythmias and/or a history of cardiovascular events including myocardial infarction, except patients with only well-controlled hypertension

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in hepatic gene expression at 45 minutes after intravenous glucose bolus compared to saline infusion | Baseline (pre-infusion, at start of surgery) to 45 minutes after infusion during bariatric surgery
  Liver biopsies are collected at two timepoints: (1) baseline, immediately after anesthesia induction and before infusion, and (2) 45 minutes after infusion of either [6,6-D2]-labeled glucose or saline. Single-cell RNA sequencing (scRNA-seq) is performed on these paired samples to measure changes in hepatic gene expression. The primary comparison is the difference in transcriptomic profiles between baseline and 45 minutes post-infusion, stratified by MASLD status (confirmed by Fibroscan and histology). Gene expression changes are quantified as fold-change in transcript abundance, normalized to baseline values.

SECONDARY OUTCOMES:
Change in gene expression in subcutaneous, omental, and visceral adipose tissue | Baseline (pre-infusion) to 45 minutes post-infusion during bariatric surgery
  Biopsies of subcutaneous, omental, and visceral adipose tissue are collected at two timepoints: (1) baseline, immediately after anesthesia induction and before infusion, and (2) 45 minutes after infusion of either [6,6-D2]-labeled glucose or saline. Single-cell RNA sequencing is performed to assess transcriptomic changes in each adipose depot. Gene expression changes are reported as fold-change relative to baseline values, stratified by MASLD status and intervention group.
Jejunal tissue gene expression profile | One-time collection during bariatric surgery
  Jejunal tissue routinely removed during Roux-en-Y gastric bypass surgery will be collected once during surgery. Transcriptomic profiling (bulk RNA sequencing) will be performed to characterize jejunal gene expression.
Plasma metabolite changes following labeled glucose infusion | Baseline (pre-infusion) to 45 minutes post-infusion during bariatric surgery
  Plasma samples collected at baseline and post-infusion will be analyzed using metabolomics to quantify changes in metabolites related to glucose catabolism, including isotope-labeled metabolites.
Insulin sensitivity index derived from IVGTT | Baseline (pre-infusion) to 45 minutes post-infusion during bariatric surgery
  Plasma glucose and insulin concentrations measured during the IVGTT will be used to calculate a prespecified insulin sensitivity index (reported as a single derived value per participant per timepoint).
Intra-jejunal microbiota composition | One-time collection during bariatric surgery.
  Intra-jejunal contents collected once during bariatric surgery will be analyzed to characterize microbiota composition.
Plasma protein changes following labeled glucose infusion | Baseline (pre-infusion) to 45 minutes post-infusion during bariatric surgery.
  Plasma samples collected at baseline and post-infusion will be analyzed using proteomic profiling to quantify changes in circulating proteins related to metabolic pathways.

CONTACTS AND LOCATIONS:
Overall Officials: Max Nieuwdorp, Prof. Dr., Principal Investigator — Amsterdam UMC
Locations (1):
- AMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided